CLINICAL TRIAL: NCT06203873
Title: A Comparison of Biodegradable and Metal Occluders in Patients With PFO and Migraine
Acronym: BioMetal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, The Vice President of Fuwai Hospital, Chinese Academy of Medical Sciences, and Director of the Structural Heart Disease Center., Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-2229
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-01

CONDITIONS: PFO - Patent Foramen Ovale; Migraine; Migraine Headache; Migraine Headache, With or Without Aura
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodegradable Occluder Cohort (Experimental)
  Interventions: Device: Biodegradable occluder
- Metal Occluder Cohort (Active Comparator)
  Interventions: Device: Metal occluder

INTERVENTIONS:
Device: Biodegradable occluder — Patients assigned in this group will receive PFO occlusion with a biodegradable occluder.
  Arms: Biodegradable Occluder Cohort
Device: Metal occluder — Patients assigned in this group will receive metal occluder for PFO occlusion
  Arms: Metal Occluder Cohort

SUMMARY:
Migraine is one of the most common chronic neurological disorders, posing a significant global public health concern. Patent Foramen Ovale (PFO) is the most common congenital heart anomaly in adults. Mechanisms linking PFO to migraine include cortical spreading depression, vascular active substance theory, impaired cerebral autoregulation, and genetic susceptibility. Understanding these mechanisms holds promise for overcoming challenges in the prevention and treatment of migraines in PFO patients. At least 11 observational studies, comprising 1,632 subjects, described the efficacy of PFO closure in cryptogenic stroke. Of these, 34% had migraines, and percutaneous PFO closure reportedly reduced migraine days by 81% (with a reduction of over 50% in monthly migraine days). Prospective randomized controlled trials (PRIMA and PREMIUM trials) assessing the Amplatzer® PFO Occluder showed significant benefits in most secondary endpoints, with a pooled analysis indicating its safety and effectiveness compared to medical therapy.While traditional metal PFO closure studies suggest symptom relief, reports also mention potential new-onset or worsened migraines post-closure. Proposed mechanisms include platelet activation, microthrombus formation, nickel allergy, and septal deformation or stretching inducing the release of migraine-related vascular active substances. However, these theories are closely tied to the presence of permanent metal implants.

Addressing these concerns, the MemoSorb® biodegradable PFO Occluder system, approved by the National Medical Products Administration (NMPA) in September 2023, offers an innovative solution. Developed collaboratively by the National Biomedical Materials Engineering Technology Research Center, Professor Wang Yunbing's team, Professor Pan Xiangbin's team from Fuwai Hospital, Chinese Academy of Medical Sciences, and HeartTech Medical, this groundbreaking technology represents a shift from metal to degradable materials. The occluder serves as a temporary bridge post-implantation, gradually degrading with endothelialization, facilitating comprehensive self-repair. This intervention concept theoretically avoids the lifelong complications associated with traditional metal occluders, effectively reducing postoperative symptoms like migraines and dizziness.

To assess and compare the treatment outcomes, especially in relieving migraines, a prospective, single-blind, randomized controlled study has been designed for patients with patent foramen ovale and migraine, comparing the novel biodegradable occluder with the metal occluder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Diagnosed migraine by ICHD-3
3. History of migraine longer than 1 year, and symptoms severely disturbing daily life.
4. TCD/TTE/TEE diagnosed patent foramen ovale with right to left shunt
5. Willing to participant and agree to follow-ups
6. Received at least three different types of migraine preventive drugs, the responder rate of previous therapy did not receive 50%.

Exclusion Criteria:

1. Migraine caused by other reason
2. Had TIA/stroke history
3. With contraindication or hypersensitive to anti-platelet or anticoagulation drugs.
4. With contraindication to PFO occlusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduced days per month at 12 month's follow-up | 12 months
  In the 12th month of follow-up, the average reduction in migraine days per month

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Z, Dong J, Dong J, Yan Y, Gao M, Fang F, Zhang F, Ouyang W, Wang S, Wang C, Pan X; BioMetal investigators. Comparison of biodegradable and metal occluders in patients with PFO and migraine: study design and rationale of BioMetal Trial. Trials. 2025 Aug 13;26(1):289. doi: 10.1186/s13063-025-09011-5. PMID 40804644